## Title: Using Facebook and Participatory Learning in an Intergenerational Intervention to Prevent Obesity in Head Start Preschoolers

IRB Approval ID: STUDY00001629

**Funding**: National Institute of Nursing Research of the National Institutes of Health under Award Number R21NR017958 (PI: Dr. Jiying Ling)

Clinical Trial Registration #: NCT04164277

Date: December 22, 2023

## PROJECT SUMMARY

Despite persistent overweight/obesity (OW/O) disparities by socioeconomic status (SES), interventions targeting preschoolers from low-SES backgrounds are sparse. Based on the intergenerational transmission of habits and obesity, targeting preschoolers and their caregivers (parents or legal guardians) simultaneously is a promising strategy for the prevention of OW/O. This project will determine the preliminary efficacy of an innovative intergenerational intervention among Head Start preschoolers, aged 3-5 years, and their caregivers. Methods: A two-group cluster randomized controlled trial will be conducted. Six Head Start centers will be randomly assigned to the intervention (n=3) or control group (n=3), and 24 caregiver-preschooler dyads will be recruited from each center (N=144 dyads). Grounded in an Actor-Partner Interdependence Model (APIM), the 16-week intervention has 3 components: 1) a caregiver component, including 1a) a Facebook-based program with weekly electronic retrievable flyers providing health information and behavioral change strategies and 4 weekly habit-formation tasks to improve parenting practices and home environment for preschoolers; and 1b) 3 face-to-face meetings (wks. 1, 8, & 16) to establish personal connections and communication networks among caregivers, discuss strategies, and share community resources to support preschoolers' behavioral changes at home; 2) a caregiver-preschooler learning component via Facebook messenger to send preschooler letters to each caregiver privately by the research team twice per week to 2a) share the preschooler's experiences of learning at school and his/her desires for a healthy diet and physical activity at home, and 2b) elicit caregivers' response to the letters; and 3) a Head Start center-based preschooler component to help preschoolers establish healthy habits via weekly healthy diet and physical activity participatory learning. AIM 1: Determine the preliminary efficacy of intervention vs control on preschoolers' proximal behavioral (e.g., MVPA, diet quality) and distal anthropometric outcomes (e.g., proportion of OW/O, BMI z-score). AIM 2: Examine the preliminary efficacy of intervention vs control on caregivers' behavioral and anthropometric outcomes. AIM 3: Compare intervention vs control on the bidirectional relationship (proposed in APIM) between preschoolers and caregivers on MVPA, diet quality, and screen time. Innovation: The intervention extends beyond prior research that focuses only on the unidirectional influence of caregivers on preschoolers with a bidirectional approach that also emphasizes the influence of preschoolers on caregivers. The potential for sustainability and scalability is high because the intervention is integrated into daily routines and capitalizes on the alreadyexisting social network Facebook to connect caregivers to an online private group. It facilitates the communication of preschooler preferences to improve caregivers' parenting practices through preschooler letters sent to caregivers via Facebook messenger. Impact: The proposed study will set the stage for a future large-scale study to prevent and reduce OW/O and promote health among underserved preschoolers.

## **PROJECT NARRATIVE**

Despite disparities in overweight/obesity (OW/O) by socioeconomic status (SES), preschoolers aged 3–5 years old from low-SES backgrounds have been underrepresented in OW/O preventive research. The proposed project, which includes low-SES caregiver-preschooler dyads and a rigorous study design, examines the preliminary efficacy of an innovative intergenerational intervention on preschoolers' proximal behavioral and distal anthropometric outcomes. This research stands to make a significant public health impact to reduce the prevalence of OW/O among underserved preschoolers, with high potential for intervention sustainability and scalability among an underserved population of concern to nursing researchers and practitioners.

**SPECIFIC AIMS**. Despite persistent disparities in overweight/obesity (OW/O) by socioeconomic status (SES), <sup>12-14</sup> and a sharp increase in obesity prevalence from 2015 (9%) to 2016 (14%) in preschoolers aged 2–5 years, <sup>15</sup> preschoolers of low SES are significantly underrepresented in OW/O preventive research. <sup>16</sup> Lifestyles promoting high-quality diet and physical activity (PA) offer the most effective approach to achieving healthy weight long-term <sup>17-19</sup> and reducing obesity-related comorbidities, <sup>20</sup> such as heart disease, <sup>21,22</sup> asthma, <sup>23</sup> impaired cognitive function, <sup>24,25</sup> metabolic syndrome, <sup>26</sup> and cancer. <sup>27</sup> Moreover, the major sociocultural root causes of OW/O in low-SES preschoolers are poor parenting practices and poor home environment. <sup>8,9,28-30</sup> Despite calls from the American Academy of Pediatrics (AAP) and the Institute of Medicine (IOM) for interventions to prevent obesity that primarily target preschoolers, <sup>31,32</sup> few interventions have been conducted with low-SES preschoolers and effects have been limited. <sup>16,33</sup> This study addresses this gap in the science in a novel manner by targeting the bidirectional participatory learning <sup>34</sup> that occurs between preschoolers and their parents or legal guardians (referred to as caregivers in this application) as an effective strategy for reducing the persistent OW/O disparities by SES<sup>35</sup> given the intergenerational transmission of health habits and obesity. <sup>36,37</sup>

Based on our prior study (n=69 dyads, see **C.2.**),<sup>38</sup> we have established the feasibility (<u>preschooler participation 77%</u>; <u>caregiver participation 87%</u>) of our 10-week, intergenerational intervention called "*FirstStep2Health.*" This intervention addresses one important root cause of OW/O—poor parenting practices —by **1)** using an existing social network, Facebook<sup>™</sup>, to involve caregivers in a private group<sup>39,40</sup> to initiate a supportive network and overcome barriers to involving working caregivers in face-to-face programs;<sup>41,42</sup> and **2)** extending the commonly used unidirectional framework of caregivers shaping preschoolers to the *bidirectional* framework—the Actor-Partner Interdependence Model (APIM)<sup>43</sup>—that adds preschoolers' preferences and how they influence caregiver-preschooler learning of healthy diet and PA.<sup>44-47</sup>

Our **long-term goal** is to promote healthy parenting practices among underserved low-SES families to reduce OW/O disparities by SES. To achieve this goal, our **16-week** (extended from 10 to 16 weeks per caregiver request in our prior study and behavior habit-formation needs 2-3 months<sup>48</sup>) **intervention** is sensitive to participants' literacy level and low-SES and includes **3 components**: **1)** a caregiver component including **1a)** a Facebook-based program with weekly electronically-retrievable flyers providing health information and behavioral change strategies and 4 weekly habit-formation tasks to create a healthier home environment for preschoolers; and **1b)** 3 face-to-face meetings (weeks 1, 8, & 16) to establish personal connections and communication networks among caregivers, discuss strategies, and share community resources to support behavioral changes at home; **2)** a caregiver-preschooler learning component<sup>34,47</sup> via Facebook messenger to send preschooler letters to each caregiver privately by the research team twice per week to share the preschooler's experiences of learning at school and his/her stated desires for healthy diet and PA at home, and to ask caregivers to respond to the letters; and **3)** a Head Start center-based preschooler component to help preschoolers establish healthy habits via weekly healthy diet and PA participatory learning.<sup>34</sup>

Our **primary objective** is to determine the preliminary efficacy of the intervention. **Methods:** We will conduct a **two-group cluster randomized controlled trial** (RCT). From the available 13 large Head Start centers, six centers will be randomly selected and then randomly assigned to the intervention (n=3) or control group (n=3, usual Head Start activities); 24 caregiver-preschooler dyads will be recruited from each center (N=144 dyads).

AIM 1: Determine the preliminary efficacy of FirstStep2Health vs control among preschoolers on proximal behavioral changes of ↑ moderate-to-vigorous PA (MVPA) measured by accelerometry (primary outcome), ↑ diet quality (e.g., ↑ fruits/vegetables, ↑ fiber, ↑ whole grains, ↑ total protein, ↑ dairy, ↓ sugarsweetened beverages, \u03c4 total sugars/fats), and \u03c4 screen time (e.g., watching TV, playing video games); and distal anthropometric outcomes of | proportion of OW/O and | body mass index (BMI) z-score. We anticipate an overall decrease in BMI z-score in intervention preschoolers because we expect OW/O preschoolers' BMI z-score to decrease and healthy-weight preschoolers to have no change. We focus on proximal behavioral changes as our primary outcome instead of distal anthropometric outcomes due to the brevity of this study and the need for behavioral changes to be maintained for at least a year before manifesting in changes in anthropometric outcomes. 49,50 AIM 2: Examine the preliminary efficacy of FirstStep2Health vs control **among caregivers** on their ↑ MVPA measured by accelerometry, ↑ diet quality (e.g., ↑fruits/vegetables, ↑fiber), ↓ screen time, ↓ proportion of OW/O, ↓ BMI, ↑ knowledge, ↑ feeding practice skill, ↑ self-efficacy, ↑ parental support of their child, ↑ parenting practices, and ↑ home environment. AIM 3: Compare FirstStep2Health vs control on the bidirectional relationship (as demonstrated in the APIM) between preschoolers and caregivers on MVPA, diet quality, and screen time. Further, we will validate established feasibility, acceptability, and satisfaction of the intervention using qualitative and quantitative data.

**Impact:** This application integrates existing best practices for preventing OW/O into an innovative intergenerational intervention that targets caregivers via existing social network Facebook™ and promotes caregiver-preschooler learning based on a bidirectional framework. This study forms the foundation for a future large-scale RCT to prevent OW/O and promote health among low-SES preschoolers.

A. SIGNIFICANCE A.1. A critical need exists to reduce overweight/obesity (OW/O) among preschoolers in low-socioeconomic status (SES) families. 13,14 About 34% of U.S. Head Start preschoolers 51,52—1.3 times the rate of U.S. children aged 2-5 years (26%)<sup>15</sup>—are OW/O. The OW/O prevalence rate was 46% in our prior study.<sup>38</sup> Disparities in OW/O by SES persist from childhood through adolescence<sup>53</sup> and are related to underlying SES disparities in dietary intake<sup>54</sup> and PA.<sup>55</sup> Children who experience poverty by 2 years of age are almost two-times more likely to be obese by age 15 compared to those not experiencing poverty at an early age. 56 Head Start programs serve children and families with incomes under the poverty thresholds. 57 **This** research is significant because it addresses the gap in literature involving studies targeting both preschoolers and their caregivers from low-SES backgrounds. 16,33,58 Intervening with preschoolers <5 yrs. old results in better short- and long-term outcomes in weight reduction compared to intervening with elementary school children (6–11 yrs.) or adolescents (≥12 yrs.). 17,18,59 Six interventions were identified that focused on low-SES Head Start preschoolers (including healthy weight and OW/O preschoolers). Two interventions used passive caregiver involvement by sending home materials, but had no effect on preschoolers' BMI.60,61 Four interventions actively involved caregivers via face-to-face classes: one resulted in a significant but small BMI decrease (d=0.17), but lacked control group and caregiver attendance data:<sup>62</sup> two had no significant BMI change with low caregiver attendance (32-38%);<sup>41,63</sup> and one used a quasi-experimental design and had a high caregiver attendance (80%), but no significant BMI change.<sup>64</sup> The high attendance may have occurred because only caregiver-transported preschoolers were included, and caregivers received the intervention when they arrived to pick up their child. Moreover, previous interventions with preschoolers only achieved a small effect on BMI (d=0.19), and the effect was even smaller (d=0.10) when including  $\geq$  50% low-SES preschoolers. 16,65 These dismal results, coupled with the sharp increase in obesity prevalence from 2015 (9%) to 2016 (14%) in preschoolers <sup>15</sup> and the low percentages of Head Start preschoolers meeting fruit/vegetable (9%)<sup>66-68</sup> and MVPA (50%)<sup>69,70</sup> recommendations, highlight the critical need for this innovative intergenerational intervention. Furthermore, health habits established in preschool years persist later in childhood,<sup>71,72</sup> highlighting the importance of introducing preventive efforts before entering kindergarten. A.2. SCIENTIFIC PREMISE. The major root causes of OW/O in low-SES preschoolers and their primary caregivers include unhealthy diet (e.g., excessive sugar drinks and fat intake, increased portion size, low intakes of fruits and vegetables), 6,73 decreased PA,6 increased screen time, 74,75 poor parenting practices, and home environment. 28-30,76 Previous interventions involving caregivers via face-to-face contact 16,33,77 resulted in low attendance (32-38%) due to inflexible caregiver schedules. 41,42,63 Internet-based interventions resulted in similar or even greater effects on weight loss compared to non-Internet-based interventions. 78-80 However, they suffer high attrition and low usage rates. 81 To address these limitations, this research uses existing social networks (i.e. Facebook)<sup>39</sup> and incorporates activities into people's daily routines.<sup>40</sup> According to the Pew Research Center, about 80% of young U.S. adults 10 and 74% of U.S. parents 11 use Facebook. In our prior study, 91% of the participating young parents used Facebook. Facebook-based interventions have achieved high retention rates (77-100%). 39,40 To date, Facebook-based interventions have focused on changing Facebook users' behaviors directly<sup>82-85</sup> but no intervention has targeted caregivers via Facebook to improve support for their preschoolers' behavioral change. Some face-to-face contact is still crucial to connect caregivers to each other to initiate a communication network<sup>86,87</sup> and create norms to boost participation.<sup>81</sup> Guided by the promising findings of our prior study, 38 we plan to extend this science in 3 ways: 1) use the existing social network Facebook<sup>™</sup> to form a private group with messaging designed to engage caregivers in the program and to create group norms to support ongoing interaction; 2) actively engage both preschoolers and their caregivers to target major root causes of OW/O including diet, PA, screen time, parenting practices, and home environment; and 3) send preschooler letters to caregivers via Facebook messenger to share their preschooler's experiences of learning at school, his/her stated desires for healthy diet and PA at home, as well as ask caregivers to provide nutritious foods and types of PA the preschooler has tried and liked. Thus, we will increase caregiver engagement and retention by forming a private homogeneous virtual community on Facebook, supplemented with limited face-to-face contact to maintain participation. Our Facebook-based program has resulted in high caregiver attendance (87%).<sup>38</sup> To our knowledge, this intervention is the first to apply a bidirectional framework that captures not only caregivers' ability to influence their preschoolers but also preschoolers' ability to influence caregivers. A bidirectional framework emphasizing the interaction between caregivers and preschoolers offers a new perspective for studying child behaviors. 88,89 Preschool is the time when a child's influence emerges. Erikson's psychosocial stage theory 90 indicates that children begin to assert autonomy by making choices about what they like between 18 months and 3 yrs. Children as young as 3 yrs. begin to have a significant role in influencing family food purchasing and consumption, 91,92 so increasing children's exposure to healthy choices will help increase their requests for

healthy items. 92 Intervening with preschoolers who begin to assert autonomy is very important to help foster an intimate, long-term, positive relationship between caregivers and children. 93-96 Prior research only emphasizes the influence of caregivers on preschoolers without considering caregiver-preschooler bidirectional influence. 45,46,97,98 Longitudinal, observational studies among preschoolers and school-age children have supported the influence of children's behaviors and weight status on parenting practices. 99-102 Experimental studies with school-age children further support that children's participation in a lifestyle intervention can significantly increase their parents' health knowledge, 103 improve home food environment, 104 and decrease parents' BMI. 105 Our study is based on the scientific promise that an intervention focusing on the bidirectional caregiver-preschooler relationship will improve behavioral and anthropometric outcomes among participants. **B. INNOVATION** This intervention is innovative because it: 1) is integrated into participants' daily routines without adding excessive burden to their daily lives to improve sustainability and scalability; 2) applies a bidirectional framework emphasizing both the influence of caregivers on preschoolers and of preschoolers on caregivers; 3) facilitates the communication of preschooler preferences to improve caregivers' feeding and activity practices through preschooler letters sent to caregivers via Facebook messenger; and 4) connects caregivers through an online private group via social network Facebook to support and motivate each other. Additionally, we apply an innovative training method to assist Head Start teachers to transition from being intervention implementation assistants to classroom education leaders: 1) MSU Extension health educators will deliver the intervention and model the role of interventionist with teachers observing for weeks 1–6; 2) Extension health educators and teachers will deliver the intervention together for weeks 7–10: 3) Teachers will deliver the intervention with Extension health educators providing on-site coaching and feedback for weeks 11–16. This training method was successful in our prior study and can help improve intervention sustainability. C. APPROACH To ensure rigor, the study will use a rigorous design, reliable and valid instruments, and training and supervision to maintain ethical conduct and intervention integrity. C.1. RESEARCH TEAM. Our multidisciplinary team includes researchers from nursing, nutrition, child

development, engineering, and biostatistics. The team includes experts in preschooler obesity prevention (PI Ling, Co-I Kerver, & Consultant Brophy-Herb), 4,38,106 Internet/social network-based intervention (PI Ling & Co-I Robbins), 38,107,108 mHealth (Co-I M. Zhang), 109-111 and cluster RCTs (Co-Is Robbins & N. Zhang). 112,113 C.2. PRELIMINARY STUDIES. In preparation for this application, we completed two systematic reviews 16,33 and two preliminary studies. 4,38,67,87 The systematic reviews 16,33 suggest that OW/O interventions should target preschoolers via participatory learning<sup>34</sup> and provide caregivers with parenting skill training and behavioral change strategies. One preliminary study,4 with 32 Head Start caregivers, identified the unique needs and barriers to healthy behaviors in Head Start families and supported the intervention strategy of involving caregivers through an online support group supplemented with face-to-face meetings. The PI collaborated with the established research team on a quasi-experimental study to examine the feasibility and preliminary efficacy of the 10-week FirstStep2Health intervention. 38,67,87 Sixty-nine dyads participated (39 in intervention). About 81% of caregivers and 46% of preschoolers were OW/O, and 92% reported no difficulty to get the foods they needed.<sup>3</sup> Feasibility. Enrollment rate was 37% and retention rate was 99%. Preschooler participation was 77%, and caregiver participation was 87%. Completion rates for weekly tasks and guizzes were 82% and 88%, respectively. About 94% of caregivers were satisfied with the program; 97% would recommend the program to others. **Efficacy.** Intervention increased MVPA (raw d=0.42) and fruit/vegetable intake (d=0.40), and decreased screen time (d=-0.21) and BMI z-score (d=-0.30) in intervention preschoolers. It also increased caregivers' fruit/vegetable intake (d=0.40), but had a small effect on their MVPA (d=0.08) and BMI (d=-0.07). Suggestions. Fifteen randomly selected caregivers were interviewed individually. They suggested: 1) holding each caregiver meeting on both weekday and weekend so working caregivers can attend; 2) covering topics on alternative cooking ingredients and portion size control during the meeting; 3) promoting more interactions via commenting on others' postings: 4) including quick meal recipes and healthy snack ideas in the intervention cookbook; and 5) extending the program a few more weeks. Results support the feasibility of the intervention, but preliminary efficacy needs further evaluation using a more rigorous design and larger sample size.



**C.3. CONCEPTUAL FRAMEWORK** (**Fig 1**). The intervention is guided by an Actor-Partner Interdependence Model (APIM),<sup>43</sup> which has been used in behavioral interventions to better understand the intergenerational relationships inside a family.<sup>114-116</sup> The APIM demonstrates the bidirectional relationship between preschoolers and caregivers: **1**) actor effects within preschoolers or caregivers, and **2**) partner effects between preschoolers and caregivers.<sup>43</sup> The proposed intervention targets both preschoolers' and caregivers' knowledge, skill, self-efficacy, and social support, derived from social cognitive theory,<sup>117</sup> and parenting practices and home environment<sup>118-123</sup> to improve their MVPA, diet quality, and screen time, thereby reducing the proportion of OW/O and BMI. Participatory learning<sup>34</sup> will be used to improve preschoolers' knowledge, skill, self-efficacy, and social support, but will not be assessed due to preschoolers' immature cognitive development.<sup>124</sup> Caregivers' learning<sup>34</sup> will be improved via weekly habit-formation tasks on child feeding practices and PA and preschooler letters where preschoolers describe their desires for healthy diet and PA at home. Through simultaneously targeting both preschoolers and caregivers to maximize the actor and partner effects, the intervention is hypothesized to result in positive outcomes.

**C.4. STUDY DESIGN**. To decrease cross-group contamination among participants in the same location, <sup>125</sup> we will employ a rigorous two-group cluster RCT design by randomizing 6 centers so participants in one center are in the same group. Data will be collected at baseline (wk. 0) and immediately post-intervention (wk. 17). **C.5. SETTING & SAMPLE**. Six Head Start centers (≥ 4 classes/center) will be randomly selected from the Capital Area Community Services (CACS) Head Start and Early Childhood Programs and the Head Start for Kent County, which had 13 centers with ≥ 4 classes in 2017. <sup>126,127</sup> Among the 13 centers, two had 4, one had 5, five had 6, one had 8, one had 9, two had 12, and one had 14 classes. The 13 centers cared for 1,932 preschoolers: 49% female, 20% Hispanic, 38% Black, and 39% White. Four classes will be randomly selected

from each center, and 6 caregiver-preschooler dyads will be randomly selected from the eligible participants in each class (total: 6 centers, 24 classes, and 144 dyads). Inclusion and exclusion criteria are specified in **Table 1**. **C.6. SAMPLE SIZE & POWER.** Due to the

C.6. SAMPLE SIZE & POWER. <u>Due to the exploratory/developmental focus of this R21 grant proposal</u>, our aim is to estimate effect sizes for proximal and distal outcomes in preschoolers to serve as foundation for future research. Assuming class cluster effects intraclass correlation (ICC)=0.01, <sup>128,129</sup> and

| Table 1. Inclusion and Exclusion Criteria | |
|---|---|
| Preschoolers | Caregivers |
| Inclusion Criteria | |
| Parental written consent | Provide written consent |
| Understand and speak English | Read, understand, and speak English |
| 3-5 years old | Primary adult caregiver (≥ 18 years old) |
| Enrolled in full-day or half-day Head | Have at least weekly Internet access |
| Start program | using a smartphone, tablet, or a computer |
| Child written assent if 5 years old | Willing to use Facebook |
| Exclusion Criteria for both | Preschoolers and Caregivers |
| Medical conditions precluding dietary changes or PA | |
| Diagnosed conditions known to impact weight (e.g., Prader-Willi Syndrome) or | |
| taking weight-affecting medications (e.g., stimulants) | |
| Diagnosed developmental disabilities | |

significance level=.05, a sample size of 130 will provide a power of .80 to identify an effect size of 0.50, < 0.66 for MVPA achieved in the prior study after adjusting for demographics.<sup>38</sup> Given the extended intervention duration from 10 to 16 weeks and the strengthened intervention, we anticipate to also achieve an effect size of 0.50 in preschoolers' diet quality, screen time, and BMI z-score. We conservatively assume a 10% dropout. C.7. RECRUITMENT. The two Head Start organizations have agreed to support implementing the proposed project in their Head Start centers (**Support Letters**). Based on our prior experiences working with Head Start families, we anticipate ≥ 6 of 18 (30%) dyads per class will be willing to participate. Replacement classes will be randomly chosen if a selected class teacher refuses to participate. Building on lessons learned from prior studies and recommendations from Head Start administrators, we will involve Head Start family advocates to help with recruitment because they already have an established, trusting relationship with each family. The PI and project manager (PM) will provide participant recruitment training with communication scripts to family advocates to ensure consistency. Family advocates will distribute the recruitment packet (including cover letter, parental consent/child assent. & screening tool) in an envelope and explain the study to each caregiver in person. Each family will be asked to return the packet in a sealed envelope to the family advocate. For nonrespondents, the family advocates will make a follow-up phone call, and then another packet will be mailed to each family. Each family will be asked to return the packet in an attached, prepaid envelope. Cash (\$5) will be provided for returning the packet. Prior to any data collection, written parental consent is required; if the child is age 5, written child assent is required. No data will be collected from preschoolers in the selected classes who do not have written consent or assent, but these preschoolers will be allowed to participate in intervention activities at their Head Start center. Both male and female preschoolers and caregivers will be recruited. C.8. RANDOMIZATION AND BLINDING. Following baseline data collection, 6 randomly selected centers will be randomly assigned to intervention or control using a computerized random-number generator. Center directors and teachers will be informed of group assignment. There is no way to completely blind participants

to group; however, having two conditions in different centers minimizes the likelihood of cross-group contamination. <sup>125</sup> Interventionists and caregivers will not be informed of the study hypothesis and will be asked not to discuss the program with others. <u>Data collectors and interviewers will be blinded to the randomization.</u> **C.9. STRATEGIES TO ENHANCE ATTENDANCE AND RETENTION.** The research team has demonstrated the ability to successfully recruit and retain participants. <sup>38,106</sup> Retention strategies include: **1)** keeping up-to-date lists of center and participant contacts; **2)** mailing thank-you cards to boost achievement following each step; **3)** using incentives to compensate for transportation and daycare cost in data collection (\$40 at baseline and \$50 post-intervention); and **4)** sending reminders via telephone calls, text messages, or emails to caregivers who have not completed data collection, weekly tasks, or logged-on to the study's Facebook group for a week. **C.10. INTERVENTION.** Rationale for the intervention duration is that 16 weeks provides a reasonable period for behavior habit formation<sup>48</sup> and is feasible for Head Start calenders. <sup>130,131</sup> Additionally, we incorporated feedback from our 10-week prior study indicating that increasing the intervention duration would be helpful. **C.10.1. Caregiver Component. Facebook-based program including 4 habit-formation tasks/wk.** (Table

2): A Facebook study site was developed in our prior study<sup>38</sup> and will be installed on each intervention caregiver's smartphone, tablet, or computer. All caregivers will be connected via a private Facebook group. We anticipate >80% will be Facebook users and >90% will have a smartphone with Internet access based

| Table 2. Caregiver Weekly Habit-Formation Tasks via Facebook | |
|---|---|
| Task | Instructions |
| Get in the | Post about a healthy meal you made for your family (e.g., make a recipe |
| kitchen | of your own OR make chicken noodle soup for your family). |
| Make active | Post about physical activity in which you helped child engage (e.g., take |
| time family time | a walk with child, play a family activity game with child). |
| Leave a positive | Positively respond to one other person's posting (e.g., Yum! That looks |
| comment | like a delicious meal. Great job.). |
| Take a quiz | Reinforce information & strategies learned (e.g., repeatedly exposing |
| | child to novel or disliked food is an effective strategy to deal with picky |
| | eaters; true or false?). |

on previous literature<sup>10,11,132</sup> and our prior study. To address the unique needs of this low-SES population,<sup>4</sup> the program will **1)** provide caregivers a weekly electronically retrievable flyer containing health information, family fun activities, and behavioral change strategies to help create a healthier home environment, and **2)** encourage interactive positive communication to promote peer support. All program materials will be sensitive to

participants' literacy level, low-SES & use of images as confirmed in our prior work. The program has 6 components (**Table 3**).

Three face-to-face caregiver meetings: MSU Extension health educators will lead the meetings at Head Start centers (wks. 1, 8, & 16; Support Letter) to connect caregivers to each other, offer health information, and discuss behavioral change strategies. To improve attendance and accommodate caregivers' work schedules, each meeting will be held on a weekday and a weekend day at each center. Healthy food

| Table 3. Caregiver Facebook-based Program Components | |
|---|---|
| Component | Contents & Instructions |
| Front Page | Caregiver progress (# tasks completed) will be updated daily on this page. |
| Complete | Each Sunday morning, caregivers will receive a notification on weekly tasks and |
| Tasks | will be asked to complete tasks by midnight the following Saturday. |
| | Each Friday morning, caregivers will receive a reminder via Facebook messenger |
| | and text messaging to complete the weekly tasks. |
| | For caregivers who have not logged-on to the study's Facebook group for a week, |
| | reminders will be sent via text message, phone call, or email aligning with their |
| | preferred communication method. |
| Past Tasks | Past tasks can still be completed after due date because some caregivers may |
| | not be able to complete on time due to illness or other personnel events. |
| | The flexibility was highly appreciated by caregivers in the prior study. |
| Take A Quiz | After completing each quiz, immediate feedback will be provided (e.g., You bet! |
| | Every minute counts. The physical activity goal of 10,000 steps/day can be |
| | achieved in sessions: a morning walk, a midday walk, and an evening walk.). |
| Encouraging | Messages on parental influence will be posted on the private Facebook group's |
| Messages | front page every other day to encourage caregivers to take little steps at a time to |
| | help make healthy behavioral changes in the family (e.g., <i>To the world, you're a</i> |
| | mother, but to your child, you are the world.). |
| Talk to a | This will allow caregivers to send private messages to the research team via |
| Researcher | Facebook messenger if needed to obtain advice on healthy diet and PA. |

taste-testing activities will be offered to expose caregivers to a variety of healthy homemade meals provided by MSU Extension. **Meeting 1**: A healthy, slow cooking demonstration will be offered, and each family will receive a small bag of groceries to facilitate preparation of the demonstrated recipe at home. Alternative cooking ingredients will be discussed to help reduce sugar and fat. Each caregiver will also receive an intervention cookbook containing affordable, slow-cooking recipes, quick-fix recipes, and healthy snack ideas. Reasons for providing a cookbook are: **1)** in our prior study, Head Start caregivers requested "quick fix," affordable but healthy, recipes; and **2)** using a slow cooker to prepare easy but healthy meals is an effective strategy to overcome low-SES parent barriers of lack of time and cooking skills. Aland Meeting **2**: Extension health educators will demonstrate how to spend less and shop healthy, and how to read nutrition fact labels to promote healthy purchasing behaviors. Each caregiver will receive two, durable plastic "MyPlate" adult and child meal-portion plates to guide their proper portion size. Meeting **3**: Extension health educators will present community healthy eating and PA resources (e.g., farmer's markets, community gardens, nearby parks or

other free or affordable PA facilities) and provide caregivers a resource manual. Each caregiver will receive a binder including all intervention materials to ensure access to intervention information after intervention ends. C.10.2. Caregiver-Preschooler Learning. Each week, preschoolers will create two letters using stickers regarding a food or activity presented in the center-based program that they liked or wanted to try at home. Letters will be sent by the PM privately to each caregiver via Facebook messenger every Wed. and Fri. Caregivers will be encouraged to discuss letters with their preschoolers and offer foods and activities desired by preschoolers. They will also be asked to answer two Facebook multiple-choice questions related to the letters each week by Sun. midnight (a. What foods listed in your child's letter did you provide? b. What activities listed in your child's letter did your family try?). Caregiver responses to the questions will be summed to indicate caregiver responses to child requests. Each preschooler's letters will be kept in his/her intervention binder with other intervention materials to present to his/her caregiver at Meeting 3. Weekly preschooler activities, with pictures or videos, will be shared with caregivers via the Facebook private group every week. C.10.3. Center-based Preschooler Component (Table 4). Built on previous research. 16,33,38,134-136 preschoolers will receive weekly, age-appropriate, participatory learning<sup>34</sup> co-delivered by teachers and MSU Extension health educators. Session duration will be 20 minutes because children's normal attention span is 3-5 minutes per year of age, 137 and 20 min/session is recommended for preschoolers.4

| Table 4. Weekly | Table 4. Weekly Healthy Eating and PA Program at Intervention Head Start Centers | | |
|---|---|---|---|
| Theme | Dose | Objectives | "Eat & Walk My ABCs" Curriculum* |
| Healthy eating learning | 20 min.<br>Mon. | Increase knowledge | <ul> <li>Learn where food comes from, how its grown, and its nutrition.</li> <li>Use food cards, costumes, food handheld puppets, and role-playing games.</li> </ul> |
| Taste-testing activities | 20 min.<br>Tues. | Expose to healthy foods | <ul> <li>Use senses to understand the foods covered on Monday (how a food looks, smells, feels, and<br/>tastes).</li> </ul> |
| Skill training | 20 min.<br>Wed. | Improve fundamental movement skill | <ul> <li>Use animal movements to teach fundamental movement skills: balance (e.g., balance on one<br/>foot, walk on a line), locomotor (e.g., running, hopping), and ball skills (e.g., kicking, throwing).</li> </ul> |
| Fun physical activity | 20 min.<br>Thur. | Increase physical activity | <ul> <li>Use fun activity games adapted from the CATCH early childhood activity box<sup>138</sup> and <i>Eat Well Play Hard</i><sup>139</sup> to practice the movement skills covered on Wednesday.</li> <li>Reflect on the benefits of participating in physical activity.</li> </ul> |

\*A nurse expert in child development, a pediatric nurse practitioner, and a Head Start dietitian reviewed and approved the curriculum.

C.11. CONTROL. Control group will receive usual Head Start activities during intervention period. After post-intervention data collection, each control caregiver will receive all intervention supplies and a mini program including a face-to-face caregiver meeting and 1-week preschooler program. The caregiver meeting will cover contents on alternative cooking ingredients, food labels, and portion sizes.

**C.12. TRAINING**. To insure intervention fidelity and high quality data, the PI, Co-Is (Robbins & Kerver), and PM will conduct an initial training on study protocol for the whole research team. MSU Extension health educators will receive additional training on the preschooler curriculum. The statistician, Dr. N. Zhang, and Co-I (Dr. M. Zhang) will also train the PM as the data manager and Facebook moderator, respectively. Training manuals will be provided to all research staff.

C.13. INTERVENTION FIDELITY MONITORING & EVALUATION. The PM will monitor the Facebook group daily to record task-completion rates and caregivers' site visits, respond to caregivers' questions and postings, and review records and posted content to ensure proper posting and functionality. Extension health educators will record caregiver meeting attendance and activities, as well as each preschooler's attendance, punctuality, participation, and activities offered for the day in a daily activity log. The PI will communicate with Extension health educators weekly to review objectives, attendance, and intervention delivery dose, and discuss issues and solutions. Head Start teachers will complete an evaluation survey on preschooler program, and caregivers will complete an evaluation survey on caregiver program and preschooler letters (Appendix A). Two process evaluators will observe 6 randomly sampled sessions (2/center; 1 session from Extension health educator and 1 session from teacher) to evaluate preschooler curriculum implementation and activity engagement. At post-intervention, individual interviews (Appendix A) with 10 randomly selected caregivers will be conducted with the PM and PI to obtain in-depth evaluation of the intervention and future suggestions for improvement.

C.14. DATA COLLECTION & OUTCOME MEASURES (Table 5, Appendix A). All outcomes will be assessed

at baseline and post-intervention. Height and weight will be measured in a private room in Head Start centers. To improve compliance with wearing accelerometers, an auto text-message reminder will be sent to caregivers every morning at 7AM via the *REDCap* web application maintained by MSU CTSI-BRIC (**Support Letter**). The 24-hour dietary recall will be administered by 4 trained interviewers via telephone<sup>140</sup> on 2 weekdays and 1 weekend day, 141,142 using the Nutrition Data System for Research (NDSR) software developed by the Nutrition Coordinating Center, 143 University of Minnesota. Trained interviewers will also observe the snacks and lunch offered at Head Start centers. Drs. Ling & Robbins, who have completed the 2-day training on NDSR, will assess and assure diet data quality. The Environment and Policy Evaluation and Observation-Self-Report (EPAO-SR) will be completed by each center supervisor and two teachers on a single day to assess each

Head Start center environment, including the physical environment, provisions, practices, policies, training, and education. All other surveys will be completed by caregivers online via REDCap web application. Caregivers will be informed of online surveys via text-message or email. Data collectors and interviewers (blinded to group assignment) will be available by phone or in-person to answer questions.

| Table 5. Study Measures | | | | |
|---|---|---|---|---|
| Concept | Measure and Description | # Items | Time | Reliability/Validity |
| Preschoolers (Aim 1) | | | | |
| MVPA (min/day) | 7-day ActiGraph GT3X-plus accelerometer <sup>145</sup> <b>Cut-points</b> : sedentary activity (≤37 counts/15 s), light (38–419), moderate (420–841), & vigorous (≥842) <sup>146,147</sup> | 7-day | 5 min | Reliability =0.69–0.84 <sup>148</sup> r =0.66 with observational system <sup>145</sup> |
| Diet quality (e.g.,<br>fruit/vegetable, fiber,<br>sugar/fat) | Intake at Head Start center: dietary observation system on snacks and lunch on two weekdays <sup>149</sup> Intake at home: proxy-reported 24-hour dietary recall | 3-day | 90 min | ICC =0.99; <sup>149</sup> accurate rate:<br>95%; <sup>150</sup> good agreement with<br>actual energy intake <sup>151</sup> |
| Screen Time | NHANES-Physical Activity and Physical Fitness survey <sup>152</sup> | 2 | 1 min | Reliability: <i>r</i> =0.63–0.84 <sup>153</sup> |
| Proportion of OW/O,<br>BMI z-score | Calculated from height and weight using CDC growth charts <sup>154</sup> <b>Height</b> : Child/Adult Shorr Measuring Board Stadiometer <b>Weight</b> : Child/Adult Seca model 874 portable electronic scale In accordance with NHANES measurement protocol <sup>155</sup> | N/A | 3 min | Specificity 0.93; sensitivity 0.73 <sup>156</sup> |
| | Caregivers (Aim 2) | | | |
| MVPA | 7-day ActiGraph GT3X-plus accelerometer <b>Cut-points</b> : light (0–2689 counts/60 s), moderate (2690–6166), & vigorous (≥6167) <sup>157</sup> | 7-day | 5 min | ICC = $0.97-0.99^{158}$<br>r = 0.81 with oxygen consumption <sup>159</sup> |
| Diet quality | Fruit-vegetable-fiber screener <sup>160</sup> | 10 | 3 min | r=0.71 with full Block survey <sup>160</sup> |
| Screen Time | NHANES-Physical Activity and Physical Fitness survey <sup>152</sup> | 2 | 1 min | Reliability: r = 0.63-0.84 <sup>153</sup> |
| Proportion of OW/O,<br>BMI | Calculated using (weight <i>kg</i> /height <i>m</i> <sup>2</sup> ) <sup>161</sup> Measures are similar to those used in preschoolers | N/A | 3 min | Specificity 0.97; sensitivity 0.42 <sup>162</sup> |
| Knowledge | Knowledge on preschoolers' dietary intake & physical activity <sup>163</sup> | 25 | 5 min | N/A |
| Feeding Practice Skill | Child Feeding Questionnaire <sup>164</sup> measuring caregiver feeding practice behaviors | 33 | 5 min | $\alpha$ =0.71-0.93 <sup>38,164,165</sup> $r$ =-0.26-0.53 with child BMI <sup>164-166</sup> |
| Self-Efficacy | Parental self-efficacy scale <sup>163</sup> | 20 | 4 min | $\alpha = 0.72 - 0.94^{38,163}$ |
| Parental Support | Parental support scale for eating habits and physical activity 167 | 12 | 3 min | $\alpha = 0.83 - 0.87^{38,167,168}$ |
| Parenting Practices | Parenting Style and Dimensions Questionnaire 169 assessing parenting styles: authoritative, authoritarian, and permissive | 32 | 5 min | $\alpha = 0.64 - 0.91^{170}$ |
| Home Environment | Family Nutrition and Physical Activity (FNPA) screening tool 171 assessing home obesogenic environments and practices | 20 | 4 min | Correlated with child BMI <sup>171,172</sup> |
| Demographics | Socio-demographic questionnaire (e.g., age, sex, race) | 12 | 3 min | N/A |
| Center Environment | EPAO-SR <sup>144</sup> | 1-day | 30 min | Related to observational data <sup>144</sup> |

C.15. DATA ANALYSIS. Any missing at random (MAR) data will be imputed using procedures suggested by Potthoff.<sup>173</sup> For non-MAR data, a sensitivity analysis will be performed following recommended approaches for continuous and discrete outcomes.<sup>174-177</sup> All analyses will use the intention-to-treat. Principle Data analysis will be disaggregated by sex in preschoolers. AIM 1 & 2: Mixed-effect models in SAS 9.4 will be used to evaluate the intervention efficacy. Fixed effect predictors will include group, time, groupXtime interaction, and potential confounders such as preschooler sex, race, baseline weight status, and caregiver marital status. The correlation of preschooler outcomes measured over time and dependence due to nesting in the same center or class will be accounted through center- and class-specific random cluster effect. Contrasts will quantify the intervention effects separately at the post-intervention. Holm's method will be used to statistically control for multiple comparisons. The effect size (Cohen's d) will be calculated. AIM 3: Path analysis will be conducted using EQS 6.2. Model fit will be assessed using root mean square error approximation, Normed Fit Index, and Tucker Lewis index. Chi-square difference test will be used to compare models. Model modification will be made if needed. Feasibility/acceptability/satisfaction will be determined through enrollment, intervention participation, and evaluation survey data. Recorded individual interviews will be analyzed using directed content analysis in ATLAS.ti 8 to evaluate reasons for satisfaction and suggestions for improvement.

| Table 6. Method Considerations | |
|---|---|
| Issue | Justification and Strategies |
| Different participation by Head Start teachers may influence intervention delivery. | <ul> <li>Based on our prior 10-wk study, all six teachers in the intervention classes independently and<br/>successfully delivered the last 4 wks. of the program.</li> </ul> |
| Compliance with wearing ActiGraphs. | <ul> <li>We will send daily auto reminders. We will replace broken or misplaced ActiGraphs. Imputation<br/>techniques will be used for missing data.</li> </ul> |
| Difficulty meeting recruitment goals. | <ul> <li>We will use Head Start family advocates to help with recruitment. Another center or class will be<br/>randomly selected if selected center or class elects not to participate.</li> </ul> |

| Table 7. Timeline for Activities | | YEAR 1 | | | YEAR 2 | |
|---|---|---|---|---|---|---|
| Months | 1-4 | 5-10 | 11-12 | 1-2 | 3-6 | 7-12 |
| IRB approval; hire/train staff; prep materials; purchase supplies. | Х | Х | | | | |
| Recruit; enroll; baseline data collection. | | Х | | | | |
| 16-week "FirstStep2Health" intergenerational intervention. | | Х | Х | X | Х | |
| Immediate post-intervention data collection. | | | | X | X | |
| Data entry, cleaning, and analysis; presentations and manuscripts. | | Х | Х | Х | Х | Х |

## REFERENCES

- 1. Burdette HL, Whitaker RC. Neighborhood playgrounds, fast food restaurants, and crime: relationships to overweight in low-income preschool children. *Prev Med.* 2004;38(1):57-63.
- 2. Burdette HL, Whitaker RC. A national study of neighborhood safety, outdoor play, television viewing, and obesity in preschool children. *Pediatrics*. 2005;116(3):657-662.
- 3. Klemetson A, Ling J. A description of food accessibility among urban head start families. The 19th Annual University Undergraduate Research and Arts Forum; 2017; Michigan State University. https://urca.msu.edu/files/forums/28/booklet/2017%20UURAF%20Program%20Book\_Digital.pdf
- 4. Ling JY, Robbins LB, Hines-Martin V. Perceived parental barriers to and strategies for supporting physical activity and healthy eating among Head Start children. *J Commun Health*. 2016;41(3):593-602.
- 5. Swinburn BA, Sacks G, Hall KD, et al. The global obesity pandemic: shaped by global drivers and local environments. *Lancet*. 2011;378(9793):804-814.
- 6. Sahoo K, Sahoo B, Choudhury AK, Sofi NY, Kumar R, Bhadoria AS. Childhood obesity: causes and consequences. *J Family Med Prim Care*. 2015;4(2):187-192.
- 7. Gurnani M, Birken C, Hamilton J. Childhood obesity: causes, consequences, and management. *Pediatr Clin North Am.* 2015;62(4):821-840.
- 8. Bates CR, Buscemi J, Nicholson LM, Cory M, Jagpal A, Bohnert AM. Links between the organization of the family home environment and child obesity: a systematic review. *Obes Rev.* 2018;19(5):716-727.
- 9. Dallacker M, Hertwig R, Mata J. The frequency of family meals and nutritional health in children: a meta-analysis. *Obes Rev.* 2018;19(5):638-653.
- 10. Smith A, Anderson M. Social media use in 2018. 2018; <a href="http://www.pewinternet.org/2018/03/01/social-media-use-in-2018/">http://www.pewinternet.org/2018/03/01/social-media-use-in-2018/</a>. Accessed April 30, 2018.
- 11. Duggan M, Lenhart A, Lampe C, Ellison NB. Parents and social media: mothers are especially likely to give and receive support on social media. 2015; <a href="http://www.pewinternet.org/2015/07/16/parents-and-social-media/">http://www.pewinternet.org/2015/07/16/parents-and-social-media/</a>. Accessed April 30, 2018.
- 12. Watts AW, Mason SM, Loth K, Larson N, Neumark-Sztainer D. Socioeconomic differences in overweight and weight-related behaviors across adolescence and young adulthood: 10-year longitudinal findings from Project EAT. *Prev Med.* 2016;87:194-199.
- 13. Bush NR, Allison AL, Miller AL, Deardorff J, Adler NE, Boyce WT. Socioeconomic disparities in childhood obesity risk: association with an oxytocin receptor polymorphism. *JAMA Pediatr.* 2017;171(1):61-67.
- 14. Tester JM, Phan TT, Tucker JM, et al. Characteristics of children 2 to 5 years of age with severe obesity. *Pediatrics*. 2018.
- 15. Skinner AC, Ravanbakht SN, Skelton JA, Perrin EM, Armstrong SC. Prevalence of obesity and severe obesity in US children, 1999-2016. *Pediatrics*. 2018.
- 16. Ling J, Robbins LB, Wen F, Zhang N. Lifestyle interventions in preschool children: a meta-analysis of effectiveness. *Am J Prev Med.* 2017;53(1):102-112.
- 17. Reinehr T, Kleber M, Lass N, Toschke AM. Body mass index patterns over 5 y in obese children motivated to participate in a 1-y lifestyle intervention: age as a predictor of long-term success. *Am J Clin Nutr.* 2010;91(5):1165-1171.
- 18. Cheng JK, Wen X, Coletti KD, Cox JE, Taveras EM. 2-Year BMI changes of children referred for multidisciplinary weight management. *Int J Pediatr.* 2014;2014:152586.
- 19. Matusik P, Malecka-Tendera E. Overweight prevention strategies in preschool children. *Int J Pediatr Obes*. 2011;6(Suppl 2):2-5.
- 20. Llewellyn A, Simmonds M, Owen CG, Woolacott N. Childhood obesity as a predictor of morbidity in adulthood: a systematic review and meta-analysis. *Obes Rev.* 2016;17(1):56-67.
- 21. Messiah SE, Arheart KL, Natale RA, Hlaing WM, Lipshultz SE, Miller TL. BMI, waist circumference, and selected cardiovascular disease risk factors among preschool-age children. *Obesity*. 2012;20(9):1942-1949.
- 22. Anderson LN, Lebovic G, Hamilton J, et al. Body Mass Index, waist circumference, and the clustering of cardiometabolic risk factors in early childhood. *Paediatr Perinat Epidemiol.* 2016;30(2):160-170.
- 23. Vijayakanthi N, Greally JM, Rastogi D. Pediatric obesity-related asthma: the role of metabolic dysregulation. *Pediatrics*. 2016;137(5).
- 24. Smith E, Hay P, Campbell L, Trollor JN. A review of the association between obesity and cognitive function across the lifespan: implications for novel approaches to prevention and treatment. *Obes Rev.* 2011;12(9):740-755.

- 25. Guxens M, Mendez MA, Julvez J, et al. Cognitive function and overweight in preschool children. *Am J Epidemiol*. 2009;170(4):438-446.
- 26. Graversen L, Sorensen TI, Petersen L, et al. Preschool weight and body mass index in relation to central obesity and metabolic syndrome in adulthood. *PLoS One.* 2014;9(3):e89986.
- 27. Arnold M, Leitzmann M, Freisling H, et al. Obesity and cancer: an update of the global impact. *Cancer Epidemiol.* 2016;41:8-15.
- 28. Musaad SMA, Speirs KE, Hayes JT, et al. The impact of environmental, parental and child factors on health-related behaviors among low-income children. *Appetite*. 2017;112:260-271.
- 29. Kaufman L, Karpati A. Understanding the sociocultural roots of childhood obesity: food practices among Latino families of Bushwick, Brooklyn. *Soc Sci Med.* 2007;64(11):2177-2188.
- 30. Jain A, Sherman SN, Chamberlin LA, Carter Y, Powers SW, Whitaker RC. Why don't low-income mothers worry about their preschoolers being overweight? *Pediatrics*. 2001;107(5):1138-1146.
- 31. Institute of Medicine. *Early childhood obesity prevention policies*. Washington, DC: The National Academies Press: 2011.
- 32. American Academy of Pediatrics. AAP updates recommendations on obesity prevention: It's never too early to begin living a healthy lifestyle. 2015; <a href="https://www.aap.org/en-us/about-the-aap/aap-press-room/pages/AAP-Updates-Recommendations-on-Obesity-Prevention-It's-Never-Too-Early-to-Begin-Living-a-Healthy-Lifestyle.aspx">https://www.aap.org/en-us/about-the-aap/aap-press-room/pages/AAP-Updates-Recommendations-on-Obesity-Prevention-It's-Never-Too-Early-to-Begin-Living-a-Healthy-Lifestyle.aspx</a>. Accessed September 22, 2017.
- 33. Ling JY, Robbins LB, Wen FJ. Interventions to prevent and manage overweight or obesity in preschool children: a systematic review. *Int J Nurs Stud.* 2016;53:270-289.
- 34. Hedges H, Cullen J. Participatory learning theories: a framework for early childhood pedagogy. *Early Child Development and Care*. 2012;182(7):921-940.
- 35. Epstein LH, Paluch RA, Wrotniak BH, et al. Cost-effectiveness of family-based group treatment for child and parental obesity. *Child Obes.* 2014;10(2):114-121.
- 36. Dolton P, Xiao M. The intergenerational transmission of body mass index across countries. *Econ Hum Biol.* 2017;24:140-152.
- 37. Haycraft E, Karasouli E, Meyer C. Maternal feeding practices and children's eating behaviours: a comparison of mothers with healthy weight versus overweight/obesity. *Appetite*. 2017;116:395-400.
- 38. Ling J, Robbins LB, Zhang N, et al. Using Facebook in a healthy lifestyle intervention: feasibility and preliminary efficacy. *Western Journal of Nursing Research*. 2018 Epub ahead of print;0(0):0193945918756870.
- 39. Maher CA, Lewis LK, Ferrar K, Marshall S, De Bourdeaudhuij I, Vandelanotte C. Are health behavior change interventions that use online social networks effective? A systematic review. *JMIR*. 2014;16(2).
- 40. Laranjo L, Arguel A, Neves AL, et al. The influence of social networking sites on health behavior change: a systematic review and meta-analysis. *J Am Med Inform Assn.* 2015;22(1):243-256.
- 41. Fitzgibbon ML, Stolley MR, Schiffer L, et al. Family-based hip-hop to health: outcome results. *Obesity*. 2013;21(2):274-283.
- 42. Lamb-Parker F, Piotrkowski CS, Baker AJL, Kessler-Sklar S, Clark B, Peay L. Understanding barriers to parent involvement in Head Start: a research-community partnership. *Early Child Res Q*. 2001;16(1):35-51.
- 43. Cook WL, Kenny DA. The actor-partner interdependence model: a model of bidirectional effects in developmental studies. *Int J Behav Dev.* 2005;29(2):101-109.
- 44. Skouteris H, McCabe M, Ricciardelli LA, et al. Parent-child interactions and obesity prevention: a systematic review of the literature. *Early Child Development and Care*. 2012;182(2):153-174.
- 45. Skouteris H, McCabe M, Swinburn B, Newgreen V, Sacher P, Chadwick P. Parental influence and obesity prevention in pre-schoolers: a systematic review of interventions. *Obes Rev.* 2011;12(5):315-328.
- 46. Ling J, Robbins LB, McCarthy VL, Speck BJ. Psychosocial determinants of physical activity in children attending afterschool programs: a path analysis. *Nurs Res.* 2015;64(3):190-199.
- 47. Baranowski T, Chen TA, O'Connor TM, et al. Predicting habits of vegetable parenting practices to facilitate the design of change programmes. *Public Health Nutr.* 2015:1-7.
- 48. Gardner B, Lally P, Wardle J. Making health habitual: the psychology of 'habit formation' and general practice. *Brit J Gen Pract*. 2012;62(605):664-666.
- 49. Hall KD, Sacks G, Chandramohan D, et al. Quantification of the effect of energy imbalance on bodyweight. *Lancet.* 2011;378(9793):826-837.

- 50. Baranowski T, Lytle L. Should the IDEFICS outcomes have been expected? *Obes Rev.* 2015;16:162-172
- 51. Aikens N, Hulsey LK, Moiduddin E, et al. *Data tables for FACES 2009 Head Start children, families, and programs: present and past data from FACES report. OPRE Report 2011-33b.* Washington, DC: Office of Planning, Research and Evaluation, Administration for Children and Families, U.S. Department of Health and Human Services; 2011.
- 52. Lumeng JC, Kaciroti N, Sturza J, et al. Changes in body mass index associated with head start participation. *Pediatrics*. 2015;135(2):e449-456.
- 53. Chen DH, Thomsen MR, Nayga RM, Bennett JL. Persistent disparities in obesity risk among public schoolchildren from childhood through adolescence. *Prev Med.* 2016;89:207-210.
- 54. Andreyeva T, Tripp AS, Schwartz MB. Dietary quality of americans by supplemental nutrition assistance program participation status a systematic review. *Am J Prev Med.* 2015;49(4):594-604.
- 55. Stalsberg R, Pedersen AV. Effects of socioeconomic status on the physical activity in adolescents: a systematic review of the evidence. *Scand J Med Sci Spor.* 2010;20(3):368-383.
- 56. Lee H, Andrew M, Gebremariam A, Lumeng JC, Lee JM. Longitudinal associations between poverty and obesity from birth through adolescence. *Am J Public Health*. 2014;104(5):E70-E76.
- 57. Head Start. Poverty guidelines and determining eligibility for participation in head start programs. 2017; <a href="https://eclkc.ohs.acf.hhs.gov/hslc/tta-system/operations/mang-sys/ersea/PovertyGuideline.htm">https://eclkc.ohs.acf.hhs.gov/hslc/tta-system/operations/mang-sys/ersea/PovertyGuideline.htm</a>. Accessed September 22, 2017.
- 58. Ward DS, Vaughn A, Story M. Expert and stakeholder consensus on priorities for obesity prevention research in early care and education settings. *Child Obes.* 2013;9(2):116-124.
- 59. Hollingworth W, Hawkins J, Lawlor DA, Brown M, Marsh T, Kipping RR. Economic evaluation of lifestyle interventions to treat overweight or obesity in children. *Int J Obesity*. 2012;36(4):559-566.
- 60. Bellows LL, Davies PL, Anderson J, Kennedy C. Effectiveness of a physical activity intervention for Head Start preschoolers: a randomized intervention study. *Am J Occup Ther.* 2013;67(1):28-36.
- 61. Davis SM, Myers OB, Cruz TH, et al. CHILE: Outcomes of a group randomized controlled trial of an intervention to prevent obesity in preschool Hispanic and American Indian children. *Prev Med.* 2016;89:162-168.
- 62. Herman A, Nelson BB, Teutsch C, Chung PJ. "Eat Healthy, Stay Active!": a coordinated intervention to improve nutrition and physical activity among Head Start parents, staff, and children. *Am J Health Promot.* 2012;27(1):e27-36.
- 63. Lumeng JC, Miller AL, Horodynski MA, et al. Improving self-regulation for obesity prevention in Head Start: a randomized controlled trial. *Pediatrics*. 2017;139(5).
- 64. Yin Z, Parra-Medina D, Cordova A, et al. Míranos! Look at Us, We Are Healthy! An environmental approach to early childhood obesity prevention. *Child Obes.* 2012;8(5):429-439.
- 65. Laws R, Campbell KJ, van der Pligt P, et al. The impact of interventions to prevent obesity or improve obesity related behaviours in children (0-5 years) from socioeconomically disadvantaged and/or indigenous families: a systematic review. *BMC Public Health*. 2014;14.
- 66. U.S. Department of Agriculture. MyPlate. 2017; <a href="https://www.choosemyplate.gov/MyPlate">https://www.choosemyplate.gov/MyPlate</a>. Accessed July 24, 2017.
- 67. Ling J, Nahry N, Wasilevich E, Robbins LB. Dietary intake among Head Start preschooler-caregiver dyads. *J Pediatr Nurs*. Under Review.
- 68. Hudson CE, Cherry DJ, Ratcliffe SJ, McClellan LC. Head Start children's lifestyle behaviors, parental perceptions of weight, and body mass index. *J Pediatr Nurs.* 2009;24(4):292-301.
- 69. Tucker P. The physical activity levels of preschool-aged children: a systematic review. *Early Child Res* Q. 2008;23(4):547-558.
- 70. Beets MW, Bornstein D, Dowda M, Pate RR. Compliance With national guidelines for physical activity in U.S. preschoolers: measurement and interpretation. *Pediatrics*. 2011;127(4):658-664.
- 71. Birch L, Savage JS, Ventura A. Influences on the development of children's eating behaviours: from infancy to adolescence. *Can J Diet Pract Res.* 2007;68(1):s1-s56.
- 72. Lytle LA, Seifert S, Greenstein J, McGovern P. How do children's eating patterns and food choices change over time? Results from a cohort study. *Am J Health Promot*. 2000;14(4):222-228.
- 73. Ebbeling CB, Pawlak DB, Ludwig DS. Childhood obesity: public-health crisis, common sense cure. *Lancet*. 2002;360(9331):473-482.
- 74. Dennison BA, Erb TA, Jenkins PL. Television viewing and television in bedroom associated with overweight risk among low-income preschool children. *Pediatrics*. 2002;109(6):1028-1035.

- 75. Mendoza JA, Zimmerman FJ, Christakis DA. Television viewing, computer use, obesity, and adiposity in US preschool children. *Int J Behav Nutr Phy.* 2007;4.
- 76. Anderson SE, Whitaker RC. Household routines and obesity in US preschool-aged children. *Pediatrics*. 2010;125(3):420-428.
- 77. Nixon CA, Moore HJ, Douthwaite W, et al. Identifying effective behavioural models and behaviour change strategies underpinning preschool- and school-based obesity prevention interventions aimed at 4-6-year-olds: a systematic review. *Obes Rev.* 2012;13 Suppl 1:106-117.
- 78. Hartmann-Boyce J, Johns DJ, Jebb SA, Aveyard P, Behavioural Weight Management Review Group. Effect of behavioural techniques and delivery mode on effectiveness of weight management: systematic review, meta-analysis and meta-regression. *Obes Rev.* 2014;15(7):598-609.
- 79. Broekhuizen K, Kroeze W, van Poppel MN, Oenema A, Brug J. A systematic review of randomized controlled trials on the effectiveness of computer-tailored physical activity and dietary behavior promotion programs: an update. *Ann Behav Med.* 2012;44(2):259-286.
- 80. Kohl LF, Crutzen R, de Vries NK. Online prevention aimed at lifestyle behaviors: a systematic review of reviews. *J Med Internet Res.* 2013;15(7):71-83.
- 81. Kelders SM, Kok RN, Ossebaard HC, Van Gemert-Pijnen JEWC. Persuasive system design does matter: a systematic review of adherence to web-based interventions. *J Med Internet Res.* 2012;14(6):17-40.
- 82. Ferrer DA, Ellis R. A review of physical activity interventions delivered via Facebook. *J Phys Act Health*. 2017:1-32.
- 83. Mendoza JA, Baker KS, Moreno MA, et al. A Fitbit and Facebook mHealth intervention for promoting physical activity among adolescent and young adult childhood cancer survivors: a pilot study. *Pediatr Blood Cancer*. 2017.
- 84. Napolitano MA, Whiteley JA, Mavredes MN, et al. Using social media to deliver weight loss programming to young adults: design and rationale for the Healthy Body Healthy U (HBHU) trial. *Contemporary Clinical Trials*. 2017;60:1-13.
- 85. Fiks AG, Gruver RS, Bishop-Gilyard CT, et al. A social media peer group for mothers to prevent obesity from infancy: the Grow2Gether randomized trial. *Child Obes.* 2017.
- 86. Vandelanotte C, Maher CA. Why we need more than just randomized controlled trials to establish the effectiveness of online social networks for health behavior change. *Am J Health Promot.* 2015;30(2):74-76
- 87. Ling J, Zahry NR, Robbins LB. Using participatory learning and parental support to assist Head Start preschoolers develop healthy habits: dose-response relationship. *Am J Health Promot*. Under review.
- 88. De Mol J, Buysse A. The phenomenology of children's influence on parents. *J Fam Ther.* 2008;30(2):163-193.
- 89. Pettit GS, Arsiwalla DD. Commentary on special section on "bidirectional parent-child relationships": the continuing evolution of dynamic, transactional models of parenting and youth behavior problems. *J Abnorm Child Psychol.* 2008;36(5):711-718.
- 90. McLeod S. Erik Érikson. 2017; <a href="http://www.simplypsychology.org/Erik-Erikson.html">http://www.simplypsychology.org/Erik-Erikson.html</a>. Accessed September 22, 2017.
- 91. Powell S, Langlands S, Dodd C. Feeding children's desires? Child and parental perceptions of food promotion to the "under 8s". *Young Consumers*. 2011;12(2):96-109.
- 92. Wingert K, Zachary DA, Fox M, Gittelsohn J, Surkan PJ. Child as change agent. The potential of children to increase healthy food purchasing. *Appetite*. 2014;81:330-336.
- 93. Kuczynski L, Parkin M. Agency and bidirectionality in socialization: interactions, transactions, and relational dialectics. In: JGrusec JE, Hastings PD, eds. *Handbook of Moral Development*. Mahwah, NJ: Erlbaum; 2006.
- 94. Clark KE, Ladd GW. Connectedness and autonomy support in parent-child relationships: links to children's socioemotional orientation and peer relationships. *Dev Psychol.* 2000;36(4):485-498.
- 95. Estrada P, Arsenio WF, Hess RD, Holloway SD. Affective quality of the mother-child-relationship longitudinal consequences for childrens school-relevant cognitive-functioning. *Dev Psychol.* 1987;23(2):210-215.
- 96. Schneider BH, Atkinson L, Tardif C. Child-parent attachment and children's peer relations: a quantitative review. *Dev Psychol.* 2001;37(1):86-100.
- 97. Pardini DA. Novel insights into longstanding theories of bidirectional parent-child influences: introduction to the special section. *J Abnorm Child Psychol.* 2008;36(5):627-631.

- 98. Byrd-Bredbenner C, Martin-Biggers J, Koenings M, Quick V, Hongu N, Worobey J. HomeStyles, a web-based childhood obesity prevention program for families with preschool children: protocol for a randomized controlled trial. *JMIR Res Protoc.* 2017;6(4):e73.
- 99. Sleddens EFC, Gubbels JS, Kremers SPJ, van der Plas E, Thijs C. Bidirectional associations between activity-related parenting practices, and child physical activity, sedentary screen-based behavior and body mass index: a longitudinal analysis. *Int J Behav Nutr Phy.* 2017;14.
- 100. Afonso L, Lopes C, Severo M, et al. Bidirectional association between parental child-feeding practices and body mass index at 4 and 7 y of age. *Am J Clin Nutr.* 2016;103(3):861-867.
- 101. Walton K, Kuczynski L, Haycraft E, Breen A, Haines J. Time to re-think picky eating?: a relational approach to understanding picky eating. *Int J Behav Nutr Phys Act.* 2017;14(1):62.
- 102. Jansen PW, de Barse LM, Jaddoe VWV, Verhulst FC, Franco OH, Tiemeier H. Bi-directional associations between child fussy eating and parents' pressure to eat: who influences whom? *Physiol Behav.* 2017;176:101-106.
- 103. Sedighi I, Nouri S, Sadrosadat T, Nemati R, Shahbazi M. Can children enhance their family's health knowledge? an infectious disease prevention program. *Iran J Pediatr.* 2012;22(4):493-498.
- 104. Heim S, Bauer KW, Stang J, Ireland M. Can a community-based intervention improve the home food environment? parental perspectives of the influence of the delicious and nutritious garden. *J Nutr Educ Behav.* 2011;43(2):130-134.
- 105. Coffield E, Nihiser AJ, Sherry B, Economos CD. Shape up somerville: change in parent body mass indexes during a child-targeted, community-based environmental change intervention. *Am J Public Health*. 2015;105(2):E83-E89.
- 106. Brophy-Herb HE, Horodynski M, Contreras D, et al. Effectiveness of differing levels of support for family meals on obesity prevention among head start preschoolers: the simply dinner study. *BMC Public Health*. 2017;17.
- 107. Hamel LM, Robbins LB. Computer- and web-based interventions to promote healthy eating among children and adolescents: a systematic review. *J Adv Nurs*. 2013;69(1):16-30.
- 108. Hamel LM, Robbins LB, Wilbur J. Computer- and web-based interventions to increase preadolescent and adolescent physical activity: a systematic review. *J Adv Nurs*. 2011;67(2):251-268.
- 109. Rahman T, Adams AT, Zhang M, et al. BodyBeat: a mobile system for sensing non-speech body sounds. Proceedings of the 12th annual international conference on Mobile systems, applications, and services: 2014: Bretton Woods, New Hampshire, USA.
- 110. Saeb S, Zhang M, Karr CJ, et al. Mobile phone sensor correlates of depressive symptom severity in daily-life behavior: an exploratory study. *J Med Internet Res.* 2015;17(7).
- 111. Zhang M, Sawchuk AA. Human daily activity recognition with sparse representation using wearable sensors. *IEEE J Biomed Health*. 2013;17(3):553-560.
- 112. Robbins LB, Pfeiffer KA, Vermeesch A, et al. "Girls on the Move" intervention protocol for increasing physical activity among low-active underserved urban girls: a group randomized trial. *BMC Public Health*. 2013;13.
- 113. Resnicow K, Zhang NH, Vaughan RD, Reddy SP, James S, Murray DM. When intraclass correlation coefficients go awry: a case study from a school-based smoking prevention study in South Africa. *Am J Public Health*. 2010;100(9):1714-1718.
- 114. Pusateri KB, Roache DJ, Kam JA. Grandparents' and young adult grandchildren's identity gaps and perceived caregiving intentions: an actor-partner interdependence model. *J Soc Pers Relat*. 2016;33(2):191-216.
- 115. Vedanthan R, Bansilal S, Soto AV, et al. Family-based approaches to cardiovascular health promotion. *J Am Coll Cardiol.* 2016;67(14):1725-1737.
- 116. Cornelius T, Desrosiers A, Kershaw T. Spread of health behaviors in young couples: how relationship power shapes relational influence. *Soc Sci Med.* 2016;165:46-55.
- 117. Bandura A. Social cognitive theory: an agentic perspective. *Annu Rev Psychol.* 2001;52:1-26.
- 118. Sallis JF, Prochaska JJ, Taylor WC. A review of correlates of physical activity of children and adolescents. *Med Sci Sport Exer.* 2000;32(5):963-975.
- 119. Sterdt E, Liersch S, Walter U. Correlates of physical activity of children and adolescents: a systematic review of reviews. *Health Educ J.* 2014;73(1):72-89.
- 120. Dolenc P, Pisot S. A review of correlates of physical activity in children and adolescents. *Didactica Slovenica-Pedagoska Obzorja*. 2010;25(2):85-96.

- 121. Pearson N, Biddle SJH, Gorely T. Family correlates of fruit and vegetable consumption in children and adolescents: a systematic review. *Public Health Nutr.* 2009;12(2):267-283.
- 122. Baranowski T, Cullen KW, Baranowski J. Psychosocial correlates of dietary intake: advancing dietary intervention. *Annu Rev Nutr.* 1999;19:17-40.
- 123. Patrick H, Nicklas TA. A review of family and social determinants of children's eating patterns and diet quality. *J Am Coll Nutr.* 2005;24(2):83-92.
- 124. Stanford Children's Health. Cognitive development. 2017; <a href="http://www.stanfordchildrens.org/en/topic/default?id=cognitive-development-90-P01594">http://www.stanfordchildrens.org/en/topic/default?id=cognitive-development-90-P01594</a>. Accessed September 22, 2017.
- 125. Donner A, Klar N. *Design and analysis of cluster randomization trials in health research.* West Sussex, United Kingdom: John Wiley & Sons, Ltd; 2000.
- 126. CACS Head Start. Capital Area Community Services (CACS), Inc. Head Start and Early Childhood Program. 2017; <a href="http://www.cacsheadstart.org/">http://www.cacsheadstart.org/</a>. Accessed August 17, 2017.
- 127. Head Start for Kent County. Annual Report 2016-2017. 2017; <a href="https://www.hs4kc.org/wp-content/uploads/2017/10/2016-2017-Annual-Report.pdf">https://www.hs4kc.org/wp-content/uploads/2017/10/2016-2017-Annual-Report.pdf</a>. Accessed March 30, 2018.
- 128. Wyatt KM, Lloyd JJ, Abraham C, et al. The Healthy Lifestyles Programme (HeLP), a novel school-based intervention to prevent obesity in school children: study protocol for a randomised controlled trial. *Trials*. 2013;14:95.
- 129. Murray DM, Catellier DJ, Hannan PJ, et al. School-level intraclass correlation for physical activity in adolescent girls. *Med Sci Sports Exerc.* 2004;36(5):876-882.
- 130. Fitzgibbon ML, Stolley MR, Schiffer L, Horn L, KauferChristoffel K, Dyer A. Hip-Hop to Health Jr. for Latino preschool children. *Obesity*. 2006;14(9):1616-1625.
- 131. Eliakim A, Nemet D, Balakirski Y, Epstein Y. The effects of nutritional-physical activity school-based intervention on fatness and fitness in preschool children. *J Pediatr Endocrinol Metab.* 2007;20(6):711-718.
- 132. Loehmer E, Smith S, McCaffrey J, Davis J. Examining internet access and social media application use for online nutrition education in SNAP-Ed participants in rural Illinois. *J Nutr Educ Behav.* 2018;50(1):75-+.
- 133. Nepper MJ, Chai W. Parents' barriers and strategies to promote healthy eating among school-age children. *Appetite*. 2016:103:157-164.
- 134. Fitzgibbon ML, Stolley MR, Schiffer LA, et al. Hip-hop to health jr. obesity prevention effectiveness trial: Postintervention results. *Obesity*. 2011;19(5):994-1003.
- 135. Davis SM, Sanders SG, FitzGerald CA, Keane PC, Canaca GF, Volker-Rector R. CHILE: an evidence-based preschool intervention for obesity prevention in Head Start. *J School Health*. 2013;83(3):223-229.
- 136. Adams J, Zask A, Dietrich U. Tooty Fruity Vegie in preschools: an obesity prevention intervention in preschools targeting children's movement skills and eating behaviours. *Health Promot J Austr.* 2009;20(2):112-119.
- 137. Chapman S. Attention problem in children: understanding attention spans of young children. 2015; http://abilitypath.org/2015/03/31/attention-problems/. Accessed September 22, 2017.
- 138. CATCH. PRE-K. 2017; http://catchinfo.org/programs/pre-k/. Accessed September 22, 2017.
- 139. New York State Department of Health. Eat Well Play Hard in child care centers. 2014; <a href="https://www.health.ny.gov/prevention/nutrition/cacfp/ewphccs.htm">https://www.health.ny.gov/prevention/nutrition/cacfp/ewphccs.htm</a>. Accessed September 22, 2017.
- 140. Tran KM, Johnson RK, Soultanakis RP, Matthews DE. In-person vs telephone-administered multiple-pass 24-hour recalls in women: validation with doubly labeled water. *J Am Diet Assoc.* 2000;100(7):777-783.
- 141. Ma YS, Olendzki BC, Pagoto SL, et al. Number of 24-hour diet recalls needed to estimate energy intake. *Ann Epidemiol.* 2009;19(8):553-559.
- 142. Hebert JR, Hurley TG, Cavicchia P, et al. Response to Dr. Arab et al on "Number of 24-hour diet recalls needed to estimate energy intake". *Ann Epidemiol.* 2010;20(1):87-88.
- 143. Schakel SF, Jasthi B, Van Heel N, Harnack L. Adjusting a nutrient database to improve calculation of percent calories from macronutrients. *J Food Compos Anal.* 2009;22:S32-S36.
- 144. Ward DS, Mazzucca S, McWilliams C, Hales D. Use of the Environment and Policy Evaluation and Observation as a Self-Report Instrument (EPAO-SR) to measure nutrition and physical activity environments in child care settings: validity and reliability evidence. *Int J Behav Nutr Phy.* 2015;12.

- 145. Van Cauwenberghe E, Gubbels J, De Bourdeaudhuij I, Cardon G. Feasibility and validity of accelerometer measurements to assess physical activity in toddlers. *Int J Behav Nutr Phys Act.* 2011;8:67.
- 146. Pate RR, Almeida MJ, McIver KL, Pfeiffer KA, Dowda M. Validation and calibration of an accelerometer in preschool children. *Obesity*. 2006;14(11):2000-2006.
- 147. Trost SG, Fees BS, Haar SJ, Murray AD, Crowe LK. Identification and validity of accelerometer cut-points for toddlers. *Obesity*. 2012;20(11):2317-2319.
- 148. Penpraze V, Reilly JJ, MacLean CM, et al. Monitoring of physical activity in young children: how much is enough? *Pediatric Exercise Science*. 2006;18(4):483-491.
- 149. Ball SC, Benjamin SE, Ward DS. Development and reliability of an observation method to assess food intake of young children in child care. *J Am Diet Assoc.* 2007;107(4):656-661.
- 150. Klesges RC, Klesges LM, Brown G, Frank GC. Validation of the 24-hour dietary recall in preschool-children. *J Am Diet Assoc.* 1987;87(10):1383-1385.
- 151. Bornhorst C, Bel-Serrat S, Pigeot I, et al. Validity of 24-h recalls in (pre-)school aged children: comparison of proxy-reported energy intakes with measured energy expenditure. *Clin Nutr.* 2014;33(1):79-84.
- 152. Centers for Disease Control and Prevention. National Health and Nutrition Examination Survey. 2017; <a href="http://www.cdc.gov/nchs/nhanes/">http://www.cdc.gov/nchs/nhanes/</a>. Accessed September 22, 2017.
- 153. Sirard JR, Bruening M, Wall MM, Eisenberg ME, Kim SK, Neumark-Sztainer D. Physical activity and screen time in adolescents and their friends. *Am J Prev Med.* 2013;44(1):48-55.
- 154. Centers for Disease Control and Prevention. About child & teen BMI. 2015; <a href="https://www.cdc.gov/healthyweight/assessing/bmi/childrens-bmi/about-childrens-bmi.html">https://www.cdc.gov/healthyweight/assessing/bmi/childrens-bmi/about-childrens-bmi.html</a>. Accessed July 20, 2017.
- 155. Centers for Disease Control and Prevention. National Health and Nutrition Examination Survey (NHANES): Anthropometry procedures manual. 2007; <a href="https://www.cdc.gov/nchs/data/nhanes/nhanes">https://www.cdc.gov/nchs/data/nhanes/nhanes</a> 07 08/manual an.pdf. Accessed August 16, 2017.
- 156. Javed A, Jumean M, Murad MH, et al. Diagnostic performance of body mass index to identify obesity as defined by body adiposity in children and adolescents: a systematic review and meta-analysis. *Pediatr Obes.* 2015;10(3):234-244.
- 157. Sasaki JE, John D, Freedson PS. Validation and comparison of ActiGraph activity monitors. *J Sci Med Sport*. 2011;14(5):411-416.
- 158. Jarrett H, Fitzgerald L, Routen AC. Interinstrument reliability of the ActiGraph GT3X+ ambulatory activity monitor during free-living conditions in adults. *J Phys Act Health*. 2015;12(3):382-387.
- 159. Kelly LA, McMillan DG, Anderson A, Fippinger M, Fillerup G, Rider J. Validity of actigraphs uniaxial and triaxial accelerometers for assessment of physical activity in adults in laboratory conditions. *BMC Med Phys.* 2013;13(1):5.
- 160. Block G, Gillespie C, Rosenbaum EH, Jenson C. A rapid food screener to assess fat and fruit and vegetable intake. *Am J Prev Med.* 2000;18(4):284-288.
- Centers for Disease Control and Prevention. About adult BMI. 2015;
   https://www.cdc.gov/healthyweight/assessing/bmi/adult\_bmi/index.html. Accessed July 20, 2017.
- 162. Okorodudu DO, Jumean MF, Montori VM, et al. Diagnostic performance of body mass index to identify obesity as defined by body adiposity: a systematic review and meta-analysis. *Int J Obesity*. 2010;34(5):791-799.
- 163. Horodynski M, Olson B, Baker S, et al. Healthy babies through infant-centered feeding protocol: an intervention targeting early childhood obesity in vulnerable populations. *BMC Public Health*. 2011:11:868.
- 164. Birch LL, Fisher JO, Grimm-Thomas K, Markey CN, Sawyer R, Johnson SL. Confirmatory factor analysis of the Child Feeding Questionnaire: a measure of parental attitudes, beliefs and practices about child feeding and obesity proneness. *Appetite*. 2001;36(3):201-210.
- 165. Corsini N, Danthiir V, Kettler L, Wilson C. Factor structure and psychometric properties of the Child Feeding Questionnaire in Australian preschool children. *Appetite*. 2008;51(3):474-481.
- 166. Anderson CB, Hughes SO, Fisher JO, Nicklas TA. Cross-cultural equivalence of feeding beliefs and practices: The psychometric properties of the child feeding questionnaire among Blacks and Hispanics. *Prev Med.* 2005;41(2):521-531.
- 167. Trost SG, Sallis JF, Pate RR, Freedson PS, Taylor WC, Dowda M. Evaluating a model of parental influence on youth physical activity. *Am J Prev Med.* 2003;25(4):277-282.

- 168. Sallis JF, Grossman RM, Pinski RB, Patterson TL, Nader PR. The development of scales to measure social support for diet and exercise behaviors. *Prev Med.* 1987;16(6):825-836.
- 169. Robinson CC, Mandleco B, Olsen SF, Hart CH. The parenting styles and dimensions questionnaire (PSDQ). In: Perlmutter BF, Touliatos J, Holden GW, eds. *Handbook of Family Measurement Techniques*. Vol 3. Thousand Oaks, CA: SAGE Publications, Inc; 2001:319-321.
- 170. Olivari MG, Tagliabue S, Confalonieri E. Parenting Style and Dimensions Questionnaire: a review of reliability and validity. *Marriage & Family Review*. 2013;49(6):465-490.
- 171. Ihmels MA, Welk GJ, Eisenmann JC, Nusser SM. Development and preliminary validation of a Family Nutrition and Physical Activity (FNPA) screening tool. *Int J Behav Nutr Phy.* 2009;6.
- 172. Ihmels MA, Welk GJ, Eisenmann JC, Nusser SM, Myers EF. Prediction of BMI change in young children with the Family Nutrition and Physical Activity (FNPA) screening tool. *Ann Behav Med.* 2009;38(1):60-68.
- 173. Potthoff RF, Tudor GE, Pieper KS, Hasselblad V. Can one assess whether missing data are missing at random in medical studies? *Stat Med Res.* 2006;15:213-234.
- 174. Daniels M, Hogan J. Reparameterizing the pattern mixture for sensitivity analysis under informative dropout. *Biometrics*. 2000;56:1241-1248.
- 175. Kaciroti N, Raghunathan TE, Schork MA, Clark NM. A Bayesian model for longitudinal count data with non-ignorable dropout. *Applied Statistics*. 2008;57:521-534.
- 176. Kaciroti N, Raghunathan TE, Schork MA, Clark NM, Gong M. A Bayesian approach for clustered longitudinal ordinal outcome with nonignorable missing data: Evaluation of an asthma education program. *J Am Stat Assoc.* 2006;101:435-446.
- 177. Kaciroti N, Schork MA, Raghunathan TE, Julius S. A Bayesian sensitivity model for intention-to-treat analysis on binary outcomes with dropouts. *Stat Med.* 2009;28:572-585.
- 178. Little R, Yau L. Intent-to-treat analysis for longitudinal studies with drop-outs. *Biometrics*. 1996;52(4):1324-1333.
- 179. Holm S. A simple sequentially rejective multiple test procedure. *Scandinavian Journal of Statistics*. 1979:65-70.
- 180. Kline RB. *Principles and practice of structural equation modelling.* 3rd ed. New York: The Guilford Press; 2011.
- 181. Flavell JH, Miller PH, Miller SA. Cognitive development. Englewood Cliffs, NJ: Prentice-Hall; 1985.
- 182. Child Welfare Information Gateway. Identification, screening, and assessment of child abuse & neglect. 2017; <a href="https://www.childwelfare.gov/topics/systemwide/assessment/family-assess/id-can/">https://www.childwelfare.gov/topics/systemwide/assessment/family-assess/id-can/</a>. Accessed April 02, 2018.
- 183. U.S. Department of Health & Human Services. Head Start program facts fiscal year 2014. 2015; <a href="https://eclkc.ohs.acf.hhs.gov/publication/head-start-program-facts-fiscal-year-2014">https://eclkc.ohs.acf.hhs.gov/publication/head-start-program-facts-fiscal-year-2014</a>. Accessed September 22, 2017.